CLINICAL TRIAL: NCT02723825
Title: A Multi Center Study of Prognostic Factors of the Distal Epiphysis of the Tibia Fracture
Brief Title: Study of Prognostic Factors of the Distal Epiphysis of the Tibia Fracture Prognosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foshan Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yueming Guo, Director, Head of Pediatric Department of Orthopedics,Clinical Professor of Guangzhou University of TCM, Foshan Hospital of Traditional Chinese Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 456074139
Record Dates: First submitted 2016-03-18; First posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Tibial Fractures; Epiphyseal Fracture
Keywords: Distal tibia; fractures; epiphyses; children
MeSH Terms: conditions — Tibial Fractures; Fractures, Bone | interventions — Closed Fracture Reduction; Open Fracture Reduction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Less or equal to 2mm (Placebo Comparator): the residual displacement is less than or equal to 2mm
  Interventions: Procedure: Closed reduction
- Between 2-4mm (Placebo Comparator): the residual shift is between 2-4mm, manual reset once again, as still between 2-4mm
  Interventions: Procedure: Closed reduction; Procedure: Open reduction
- Greater than 4mm (Active Comparator): the residual displacement is greater than 4mm
  Interventions: Procedure: Open reduction

INTERVENTIONS:
Procedure: Closed reduction — Treated with Manipulatio, using plywood, gypsum or external fixation support to fixed
  Other Names: Manipulative reduction and External fixation
  Arms: Between 2-4mm; Less or equal to 2mm
Procedure: Open reduction — Open reduction and internal fixation
  Arms: Between 2-4mm; Greater than 4mm

SUMMARY:
Background: Epiphysis of distal end of tibia fracture is quite common in children epiphysis injury, because of the complex damage mechanism and often leads to growth retardation and joint deformity, the patient's physical and mental damage larger; also epiphysis injury restoration requires higher standard and more difficult to fixed, and methods are being actively explored to improve the curative effect and prevent the sequelae. Our hospital pediatric department of orthopedics expects to conduct prospective study through multi center to study the influence of factors such as the tibia epiphysis fracture of distal injury's mechanism and initial and residual displacement and treatment etc. on patients' prognosis of late growth disorders, joint deformity and ankle function.

Methods and analysis: To join the multi center research collaboration group of the south pediatric department of orthopedics (including Pediatric Department of orthopedics of Wuhan Union Hospital, Wuhan Tongji Hospital, Hunan Children's Hospital, Wuhan women and children's Hospital, Foshan Hospital of traditional Chinese medicine, Shenzhen children's Hospital, Guangzhou city women and children's Medical Center), the formation of multi center research network, writing program, including the inclusion and exclusion criteria, grouping and follow-up time, method. Participating in the working group meeting, listening to the expert's opinions to improve research programs, formulate the tracking table of distal tibial epiphyseal fracture, and starting to implement after approved by the medical ethics committee of each hospital. The hospital is responsible for supervision in the whole process of project implementation, and building the real-time reporting system, and it is the responsible person of pediatric department of orthopedics of Foshan Hospital of TCM to do the random inspection. After the completion of data collection, data entry and statistical analysis conducted by the pediatric department of orthopedics in Foshan Hospital of TCM.

Ethics and promotion: The research is approved by the hospital medical ethics committee of the south pediatric orthopedics multi center cooperative research group. Single blind method is performed for children in the course of the study. Research data is shared by all participating units and joints promotion of research results.

Registration: To register and update the study on the United States NIH ClinicalTrials.gov website.

DETAILED DESCRIPTION:
Introduction Epiphyseal and Epiphyseal plate are all immature skeletal growth mechanism, the epiphyseal plate injury also known as epiphyseal injuries, fracture line through the epiphyseal plate can also spread to the epiphysis or metaphysis. Epiphyseal plate's connection is weaker than normal tendon, ligament, or joint capsule, so the children of epiphyseal injuries are common. Distal tibial epiphyseal injuries accounted for about 25%- 38% of the epiphyseal injuries. Because after the injury of the distal epiphysis of the tibia injury often leads to growth retardation and joint deformity, the patient's physical and mental damage larger. Because of the complexity of the pathogenesis of this disease, and there are many related factors. The research of related factors of the disease is benefit to evaluate the prognosis, and conducive to early intervention, benefit to avoid the occurrence or development of severe sequelae, has positive significance in clinical practice.

Because the disease is related to many factors, and the serious cases of this disease are less, the multi center cooperation is conducive to the collection of sufficient cases to analyze and achieve the objective and effective results, so establish the multi center topic.

Design and overview In epiphyseal growth stage, the epiphyseal plate connects weaker than normal tendons, ligaments, or joint capsule, so epiphyseal plate is more vulnerable to be injured. Every epiphyseal complex is composed of each epiphysis and epiphyseal plate, its growth and blood supply are interdependent, which any damage may reinforce each other. The Ranvier district around the epiphysis has the ability to ossify. It is easy to form a bone bridge and growth arrest and angular deformity after injury. Epiphyseal fracture is belongs to intra-articular fractures, such as not timely reset, prone to complications. About 15% of children with fractures involving the epiphyseal injuries, the number of boys are more than girls, as the chance of injury is more, this is because men's epiphyseal plate closure time later than women's. X-ray manifestation of epiphyseal injuries, while more complex, but the epiphyseal and backbone of the corresponding position of the dislocation and epiphyseal line broadening is the most important, a slight shift and (or) epiphyseal line broadening is the most easy to be ignored, should X-ray the healthy side at the same time.

In theory, fracture involving the epiphyseal growth plate and articular surface is easily occurred in two kinds of complications: first distal tibia epiphyseal premature closure causes valgus or varus malleolus and limb shortening; the second is the distal tibial articular surface damage causes the ankle joint degenerative changes and bone arthritis. According to Salter Harris bone epiphysis injury types were divided into five types, and in the distal tibial epiphysis injury I, II type are common in clinic. Therefore, the biggest problem is the formation of the bone bridge, early epiphyseal closure, resulting in growth arrest, angular deformity. From the current literature, the most important related factors are in injured mechanism and degree of displacement Leary JT's research shows: the initial fracture displacement and damage mechanism for determining development of PPC after the fracture of epiphysis of distal end of tibia may have a significant predictive value. Ankle fracture Lauge - Hansen parting is ankle fracture classification system put forward by Lauge - Hansen doctors in 1950 according to the damage position and violence that cause deformity, able to quickly assess the damage mechanism of 90% - 95% cases, and has been widely used. Its clinical significance lies in: 1 find fracture and classify injury and be able to make the diagnosis of ligament injury. 2 guide manipulative reduction. The general principle is: closed manipulative reduction and fracture have the opposite force mechanism.3 for the distal tibial epiphysis fracture, can also understand the severity of the injury and the existence of the risk of soft tissue embedded. Therefore, we think, it is necessary to research on the lauge Hansen classification and correlation of prognosis. The relationship between the fracture displacement and correlation of prognosis is in the extent of the shift, the vast majority of doctors think less than 2mm shift can be accepted, and to shift more than 2mm, there are different opinions. Gonc U et al think ankle joint fracture usually involving the tibia and fibular epiphyses in children and adolescents. Although they do not occur with growth arrest, but may still lead to traumatic arthritis. Therefore, for more than 2 mm of residual displacement there is a need for surgical treatment. And David podeszwa Da thinks is greater than 3mm residual displacement often means embedded with soft tissue, may increase early closure of epiphysis of probability. Russo F the most pessimistic, he thinks a shift of the S - H type Ⅱ tibial distal epiphyseal fracture is a challenging problem. Rate of epiphyseal early closure is very high (> 43%). Even if incision and anatomical repositioning, removal of embedded organization, also cannot reduce the incidence of PPC, and may increase the risk of subsequent surgery.

Considered in the design, what JOHN A.O GDEN points out "epiphyseal separation should be reset as soon as possible, each delay 1 d will increase the difficulty as it repair soon. For type II epiphyseal injuries after more than 10 d, if you don't use excessive force can not make manual reduction success, however it could damage the cartilage epiphyseal plate and damage the early osteotylus, therefore, for type II epiphyseal injuries that see a doctor later (after (7-10 d) ,had better let it be malunion, and cannot use powerful technique or surgical repositioning, lest cause obvious epiphyseal growth stopped, heals the residual deformities can then use the appropriate correction osteotomy". This view is widely agreed. In the inclusion criteria we chose cases that injury within 7 days. In addition, the Risser ilium epiphyseal ossification sign is a commonly used method for determination of the bone age, JiShiJun's pediatric bone science thinks " ossification of the crista iliaca is usually in conformity with the stop of limbs' longitudinal growth", this is the important index for determining growth potential in include and exclude criteria in this topic, so there is reason to believe that when a Risser sign V degrees distal tibial epiphyseal growth stopped, fixed limb length and Angle.

Grouping Divide the patients into groups according to the residual displacement of the fracture after the first manual reduction.

Group A: the residual displacement is less than or equal to 2mm, select closed reduction and external fixation (such as splint, plaster or traction, frame of external fixation, etc.) Group B: the residual shift is between 2-4mm, manual reset once again, as still between 2-4mm, the cooperation of each unit to choose closed reduction.

Group C: the residual shift is between 2-4mm, manual reset once again, as still between 2-4mm, the cooperation of each unit to choose closed reduction.

Group D: residual displacement is greater than 4mm, open reduction and internal fixation.

Evaluation criteria According to OVADIA et al' evaluation criteria: excellent, Joint function restore basic consistent with that of the healthy side, without any symptoms, or joint flexion range is more than 75% of the healthy side, mild sore and swollen after walking, restore normal work; Good, joint flexion range is 50% - 70% of the healthy side, joint is mild soreness, markedly swollen after walking, unable to attend the heavy physical work; Can, joint flexion range is 25% - 50% of the healthy side, joint is obvious swelling and pain, difficulty walking, and accept joint arthrodesis at the end; Poor, joint range is less than 25% of the healthy side, joint is markedly swollen, pain, stiffness, unable to walk, and accept joint arthrodesis at the end.

Data collection To hospital after conventional laboratory tests, X-ray the anteroposterior and lateral film of the affected side, the contralateral tibiofibula (including ankle) and posteroanterior radiograph of pelvis, scan the affected ankle with CT (fracture displacement measurement, tibial epiphyseal radius vector and the transverse diameter and cross section). Select cases according to the inclusion criteria, exclusion criteria Divide the patients into groups according to the X-ray films of the affected side, the degree of displacement after measuring residual displacement after the first manual reduction.

Treated according to the grouping, 3 months, 6 months, 9 months, 1-5 years after surgery follow-up.Between 3 to 12 months, each time X-ray films were taken on both ankles, observe whether there are the early closure of epiphysis; 1 to 5 years, each time we measure whether the tibia shortening or angle, OVADIA efficacy assessment and ankle function evaluation (using the table of "AOFAS Ankle-Hindfoot Scale "), until 5 years long and the distal tibial epiphyseal closure of the other side.

Organization and implementation The projects will be written by Foshan Hospital of TCM pediatric orthopaedic and submitted to the south pediatric orthopaedic multicenter study group. The project design will be discussed, modified by the hospital experts. The projects will be submitted for approval by the hospital medical ethics committee. Then the various units sign a cooperation agreement after the experts determine and clear scientific, the feasibility of this topic, and the study will be registered on the United States NIH ClinicalTrials.gov website and updated according to the situation.

In the process of implementation, the southern pediatric orthopaedic multicenter study group will communicate and consult with each other to timely solve the problems and difficulties appeared in the research through the email, WeChat and phone, even on a business trip and other means of collaboration, besides the plenary meeting each quarter, to ensure the implementation of this project.

Data collection and management Statistic analysis Foshan Hospital of TCM pediatric orthopaedic formulated the tibial distal epiphyseal fracture tracking table and send it every cooperative unit to record whether there is patients epiphyseal closed early, and if there is, record the shortening length of the affected limb and angle of angulation deformity, and record the ankle limb function (valgus, varus and back stretch, plantar flexion), assess the pain index and rank according to the evaluation criteria of OVADIA etc. During the implementation of the project, the data should be filled in the table timely, accurately and objectively by cooperative unit, to keep a record of each item shall be seriously not omissions, and regular follow-up. At the same time, set up the monitor, regularly or randomly go to the test center to check and ensure that the original data is real and effective. Accounting personnel chose by Foshan Hospital of TCM to do the double entry, ensure the data entry is correct. If in doubt, the monitor will investigate then return the data. Use the SPSS16.0 to input the data, and describe normal measurement data with mean + / - standard deviation, average between the group by t test, counting data, with chi-square, finally with Logistic regression model to analysis multi-factor.

ELIGIBILITY:
Inclusion Criteria:

* The fresh fractures, within 7 days
* Closed fracture
* Type S-H I or II
* Unilateral limb fracture, no other parts of the fractures or damage
* On the other side of the lower extremity was normal
* Epiphysis is not closed and Risser sign 0-IV degrees
* No metabolic, genetic sex diseases etc.
* Signed informed consent

Exclusion Criteria:

* Old fracture, more than 8 days.
* Open injury
* Type S-H III or IV or V
* Multiple fractures and injuries
* The contralateral limb was abnormal
* Epiphyseal closure or Risser sign V degree
* There are metabolic or genetic diseases
* Do not agree to sign informed consent, not on time to follow-up.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2016-03; Primary Completion 2021-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation criteria of OVADIA and the change over time | 1 year,2year,3year,4year,5year(We think that develops gradually of limb shortening or angle because of early epiphyseal closure will result in a lowered grad of OVADIA)
  Excellent, Joint function restore basic consistent with that of the healthy side, without any symptoms, or joint flexion range is more than 75% of the healthy side, mild sore and swollen after walking, restore normal work; Good, joint flexion range is 50% - 70% of the healthy side, joint is mild soreness, markedly swollen after walking, unable to attend the heavy physical work; Can, joint flexion range is 25% - 50% of the healthy side, joint is obvious swelling and pain, difficulty walking, and accept joint arthrodesis at the end; Poor, joint range is less than 25% of the healthy side, joint is markedly swollen, pain, stiffness, unable to walk, and accept joint arthrodesis at the end.

SECONDARY OUTCOMES:
Early closure of epiphysis | 3 months，6 months,9months,12months
  Yes/No
Limb shortening | 1 year,2year,3year,4year,5year
  The length difference between the two tibia
Ankle joint function and the change over time | 1 year,2year,3year,4year,5year(We think that develops gradually of limb shortening or angle because of early epiphyseal closure will also result in a lower score of AOFAS Ankle-Hindfoot Scale)
  Use AOFAS Ankle-Hindfoot Scale to score

CONTACTS AND LOCATIONS:
Overall Officials: Yueming Guo, benco, Study Chair — Director of pediatric orthopaedic

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Russo F, Moor MA, Mubarak SJ, Pennock AT. Salter-Harris II fractures of the distal tibia: does surgical management reduce the risk of premature physeal closure? J Pediatr Orthop. 2013 Jul-Aug;33(5):524-9. doi: 10.1097/BPO.0b013e3182880279. PMID 23752150
- [Background] Leary JT, Handling M, Talerico M, Yong L, Bowe JA. Physeal fractures of the distal tibia: predictive factors of premature physeal closure and growth arrest. J Pediatr Orthop. 2009 Jun;29(4):356-61. doi: 10.1097/BPO.0b013e3181a6bfe8. PMID 19461377
- [Result] Podeszwa DA, Mubarak SJ. Physeal fractures of the distal tibia and fibula (Salter-Harris Type I, II, III, and IV fractures). J Pediatr Orthop. 2012 Jun;32 Suppl 1:S62-8. doi: 10.1097/BPO.0b013e318254c7e5. PMID 22588106
- [Result] Gonc U, Kayaalp A. [Ankle fractures in children and adolescents]. Acta Orthop Traumatol Turc. 2004;38 Suppl 1:127-37. Turkish. PMID 15187469